CLINICAL TRIAL: NCT01052714
Title: Management of Antipsychotic Medication Associated Obesity - 2
Brief Title: Healthy Lifestyles for Mentally Ill People Who Have Experienced Weight Gain From Their Antipsychotic Medications - 2
Acronym: MAMAO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D7358-R
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2017-10-06 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Diabetes; Obesity; Weight Gain
Keywords: Antipsychotic; Bipolar; Diabetes; Mental Illness; Nutrition; Obesity; Schizoaffective; Schizophrenia; Weight Gain; Weight Loss
MeSH Terms: conditions — Diabetes Mellitus; Obesity; Weight Gain; Mental Disorders; Schizophrenia; Weight Loss

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Usual Care (No Intervention): Control group with time-matched study visits
- Lifestyle Balance (Active Comparator): Weight management group education and individual counseling
  Interventions: Behavioral: Lifestyle Balance
- Usual Care then Lifestyle Balance (Other): Participants originally randomized to Usual Care, allowed to change over to Lifestyle Balance at month 6 per their request.
  Interventions: Behavioral: Lifestyle Balance

INTERVENTIONS:
Behavioral: Lifestyle Balance — Patients assigned to the behavioral weight loss program (Lifestyle Balance Program) will do the following: -Meet with their psychiatrist and a nutritionist who will go over diet recommendations with the patient - Be given a 7% weight loss goal - Be assisted in obtaining a 500 calorie reduction per day -Exercise for at least 30 min/day, at least 5 days a week - Maintain weekly food and exercise diaries -Be quizzed on their knowledge of healthy eating habits and nutrition
  Other Names: Lifestyle Balance Program
  Arms: Lifestyle Balance; Usual Care then Lifestyle Balance

SUMMARY:
This program aims to help Veterans who take antipsychotic medications lose weight. We use a program based on the American Diabetes Association's "Diabetes Prevention Program," and we have modified it to fit the lifestyles of people with mental illness. All participants are educated about nutrition and cutting down fat intake, how and when to exercise, and the causes of diabetes and how to prevent it. Participants must be Veterans who live within one hour of the Long Beach, West Los Angeles, Sepulveda, or West Los Angeles VA hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran
* Diagnosis of psychotic disorders, schizophrenia, schizoaffective disorder and bipolar illness
* Age 18-70
* Clinically determined to require ongoing treatment with Second Generation Antipsychotics (SGA) such as olanzapine, risperidone, quetiapine, ziprasidone, aripiprazole, clozapine
* Experienced weight gain since treatment with SGA's
* Inpatient or outpatient at Long Beach, West Los Angeles, Sepulveda, or Downtown VA
* Competent to sign informed consent

Exclusion Criteria:

* Have recently been diagnosed with schizophrenia (less than 1 year)
* Are pregnant or breast feeding a baby
* Have a medically unstable condition

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2015-05-28 (Actual); Study Completion 2015-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donna Ames, MD, Principal Investigator — VA Greater Los Angeles Healthcare System, West Los Angeles, CA
Locations (3):
- United States (3):
  - VA Long Beach Healthcare System, Long Beach, CA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, Sepulveda, CA, Sepulveda, California
  - VA Greater Los Angeles Healthcare System, West Los Angeles, CA, West Los Angeles, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwan CL, Gelberg HAL, Rosen JA, Chamberlin V, Shah C, Nguyen C, Pierre JM, Erickson ZD, Mena SJ, King M Jr, Arnold I, Baker MR, Meyer HB, Ames D. Nutritional counseling for adults with severe mental illness: key lessons learned. J Acad Nutr Diet. 2014 Mar;114(3):369-374. doi: 10.1016/j.jand.2013.12.005. No abstract available. PMID 24534370
- [Background] Gelberg HA, Kwan CL, Mena SJ, Erickson ZD, Baker MR, Chamberlin V, Nguyen C, Rosen JA, Shah C, Ames D. Meal replacements as a weight loss tool in a population with severe mental illness. Eat Behav. 2015 Dec;19:61-4. doi: 10.1016/j.eatbeh.2015.06.009. Epub 2015 Jul 2. PMID 26172565
- [Result] Erickson ZD, Kwan CL, Gelberg HA, Arnold IY, Chamberlin V, Rosen JA, Shah C, Nguyen CT, Hellemann G, Aragaki DR, Kunkel CF, Lewis MM, Sachinvala N, Sonza PA, Pierre JM, Ames D. A Randomized, Controlled Multisite Study of Behavioral Interventions for Veterans with Mental Illness and Antipsychotic Medication-Associated Obesity. J Gen Intern Med. 2017 Apr;32(Suppl 1):32-39. doi: 10.1007/s11606-016-3960-3. PMID 28271424
- [Derived] Tessier JM, Erickson ZD, Meyer HB, Baker MR, Gelberg HA, Arnold IY, Kwan C, Chamberlin V, Rosen JA, Shah C, Hellemann G, Lewis MM, Nguyen C, Sachinvala N, Amrami B, Pierre JM, Ames D. Therapeutic Lifestyle Changes: Impact on Weight, Quality of Life, and Psychiatric Symptoms in Veterans With Mental Illness. Mil Med. 2017 Sep;182(9):e1738-e1744. doi: 10.7205/MILMED-D-16-00405. PMID 28885930

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from outpatient mental health clinics at four southern California VA facilities occurred from September 2010 through March 2014.
Pre-assignment Details: Participants were terminated from study prior to randomization to study groups due to screen failure or withdrawal from study during the baseline assessment period.
Groups:
- Lifestyle Balance: Weight management group education and individual counseling
  Patients randomized to the Lifestyle Balance Program will do the following:
  * Meet with their psychiatrist and a nutritionist who will go over diet recommendations with the patient
  * Be given a 7% weight loss goal
  * Be assisted in obtaining a 500 calorie reduction per day
  * Exercise for at least 30 min/day, at least 5 days a week
  * Maintain weekly food and exercise diaries
  * Be quizzed on their knowledge of healthy eating habits and nutrition
- Usual Care Then Lifestyle Balance: Participants originally randomized to Usual Care, allowed to change over to Lifestyle Balance at month 6 per their request.
  Patients randomized to the Lifestyle Balance Program will do the following:
  * Meet with their psychiatrist and a nutritionist who will go over diet recommendations with the patient
  * Be given a 7% weight loss goal
  * Be assisted in obtaining a 500 calorie reduction per day
  * Exercise for at least 30 min/day, at least 5 days a week
  * Maintain weekly food and exercise diaries
  * Be quizzed on their knowledge of healthy eating habits and nutrition
Period: Overall Study
Arm/Group | Usual Care | Lifestyle Balance | Usual Care Then Lifestyle Balance
Started | 42 | 62 | 17
Completed | 17 | 33 | 15
Not Completed | 25 | 29 | 2
Not completed — Adverse Event | 6 | 3 | 0
Not completed — Death | 1 | 2 | 0
Not completed — Lost to Follow-up | 2 | 3 | 0
Not completed — Physician Decision | 9 | 9 | 1
Not completed — Withdrawal by Subject | 7 | 12 | 1

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Control group with time-matched study visits
  Includes 17 participants who would later join "Usual Care then Lifestyle Balance" group to receive the Lifestyle Balance intervention.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Lifestyle Balance | Total
Number analyzed (Participants) | 59 | 62 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 58 | 61 | 119
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.54 (10.0) | 51.87 (9.3) | 51.22 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 27
  Male | 42 | 52 | 94
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American or Black | 19 | 19 | 38
  Asian or Pacific Islander | 3 | 2 | 5
  Caucasian, White | 22 | 31 | 53
  Hispanic, Latino, or Spanish Origin | 8 | 8 | 16
  Native American or Alaska Native | 3 | 1 | 4
  Mixed Heritage or Other | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 59 | 62 | 121
Living Situation [Count of Participants; unit: Participants] — Self-selected description of living situation. Population: One Usual Care subject declined to respond.
  Participants
    Own Home: number analyzed (Participants) | 58 | 62 | 120
    Own Home | 2 | 11 | 13
    Rental Home/Apt: number analyzed (Participants) | 58 | 62 | 120
    Rental Home/Apt | 26 | 23 | 49
    With Relatives: number analyzed (Participants) | 58 | 62 | 120
    With Relatives | 10 | 11 | 21
    Board and Care: number analyzed (Participants) | 58 | 62 | 120
    Board and Care | 17 | 16 | 33
    Transitional: number analyzed (Participants) | 58 | 62 | 120
    Transitional | 3 | 1 | 4
Education [Count of Participants; unit: Participants] — Self-selected description of highest education level reached. Population: One Usual Care subject declined to respond.
  Participants
    No diploma: number analyzed (Participants) | 58 | 62 | 120
    No diploma | 2 | 3 | 5
    High School Diploma/GED: number analyzed (Participants) | 58 | 62 | 120
    High School Diploma/GED | 49 | 47 | 96
    Bachelor's or Equivalent Degree: number analyzed (Participants) | 58 | 62 | 120
    Bachelor's or Equivalent Degree | 6 | 10 | 16
    Higher Prof. Degree: number analyzed (Participants) | 58 | 62 | 120
    Higher Prof. Degree | 1 | 2 | 3
Marital Status [Count of Participants; unit: Participants]
  Married | 5 | 12 | 17
  Single/Cohabiting | 28 | 33 | 61
  Divorced/Widower | 26 | 17 | 43
Job Status [Count of Participants; unit: Participants] — Self-selected description of employment situation. Unpaid=homemaker, student, volunteer; None=retired, disabled. Population: One Usual Care and one Lifestyle Balance subject declined to respond.
  Participants
    Paid Work: number analyzed (Participants) | 58 | 61 | 119
    Paid Work | 3 | 9 | 12
    Unpaid Work: number analyzed (Participants) | 58 | 61 | 119
    Unpaid Work | 7 | 8 | 15
    None: number analyzed (Participants) | 58 | 61 | 119
    None | 48 | 44 | 92
Diagnosis [Count of Participants; unit: Participants] — Based on Diagnostic and Statistical Manual-IV criteria
  Participants
    Schizophrenia | 21 | 19 | 40
    Schizoaffective | 13 | 22 | 35
    Bipolar | 12 | 5 | 17
    Multiple | 7 | 10 | 17
    Other | 6 | 6 | 12
Antipsychotic (Weight Gain Risk) [Count of Participants; unit: Participants] — Seven Usual Care and seven Lifestyle Balance participants were documented to be on Multiple antipsychotic medications. They are reported in the "Multiple" category, and also contribute to the tally of each of those antipsychotic medications.
  Participants
    Olanzapine/Clozapine (High) | 9 | 8 | 17
    Risperidone/Quetiapine (Med) | 30 | 30 | 60
    Aripiprazole/Ziprasidone (Low) | 22 | 24 | 46
    Other | 5 | 7 | 12
    Multiple | 7 | 7 | 14
Length of Illness [Mean (Standard Deviation); unit: years] | 21.40 (13.1) | 21.46 (14.0) | 21.43 (13.5)
Age at Onset [Mean (Standard Deviation); unit: years] | 29.07 (10.4) | 30.11 (12.8) | 29.58 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Weight Change Per Week From Baseline to Termination
Description: Participants' weight was measured at each visit by study personnel using hospital scales, and the study groups' average weight changes per week were compared.
Time Frame: Up to 19 observations per person, weekly for the first 2 months, then monthly for 10 months.
Population: Analysis excludes 17 Usual Care participants who would later self-select (breaking their randomization) to join "Usual Care then Lifestyle Balance" group to receive the Lifestyle Balance intervention.
Measure: Mean (Standard Error); unit: Pounds per week
Groups:
- Lifestyle Balance: Weight management group education and individual counseling to review goals and diet and exercise journals.
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Pounds per week | 0.133 (0.057) | -0.0756 (0.0135)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p < .001, Mixed Models Analysis

2. Primary Outcome: Mean Waist Circumference Change Per Week From Baseline to Termination
Description: Participants' waist circumference was measured at each visit by study personnel using a measuring tape, and the study groups' average waist circumference changes per week were compared.
Time Frame: Up to 19 observations per person, weekly for the first 2 months, then monthly for 10 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Inches per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Inches per week | -0.011 (0.0136) | -0.016 (0.003)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.718, Mixed Models Analysis

3. Primary Outcome: Mean Body Mass Index (BMI) Change Per Week From Baseline to Termination
Description: Study personnel calculated each participant's BMI at each visit using their weight measurement taken at that visit and their height measurement taken at baseline. The study groups' average BMI changes per week were then compared.
Time Frame: Up to 19 observations per person, weekly for the first 2 months, then monthly for 10 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Units on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Units on a scale per week | 0.035 (0.011) | -0.009 (0.002)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p < .001, Mixed Models Analysis

4. Primary Outcome: Mean Serum Insulin Level Change Per Week From Baseline to Termination
Description: Results obtained through VA facility's Outpatient Lab. The study groups' average serum level changes per week were then compared.
Time Frame: Up to 5 observations per person, at baseline, 3 months, 6 months, 9 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Pmol/L per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Pmol/L per week | -0.018 (1.23) | -0.44 (0.28)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.676, Mixed Models Analysis

5. Primary Outcome: Mean Triglycerides Level Change Per Week From Baseline to Termination
Description: Results obtained through VA facility's Outpatient Lab. The study groups' average blood level changes per week were then compared.
Time Frame: Up to 5 observations per person, at baseline, 3 months, 6 months, 9 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Mg/dL per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Mg/dL per week | 5.13 (2.31) | -0.2 (0.45)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.141, Mixed Models Analysis

6. Primary Outcome: Mean Low-Density Lipoprotein (LDL) Cholesterol Level Change Per Week From Baseline to Termination
Description: as for outcome 5
Time Frame: Up to 5 observations per person, at baseline, 3 months, 6 months, 9 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Mg/dL per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Mg/dL per week | -0.031 (0.105) | 0.218 (0.208)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.92, Mixed Models Analysis

7. Primary Outcome: Mean High-Density Lipoprotein (HDL) Cholesterol Level Change Per Week From Baseline to Termination
Description: as for outcome 5
Time Frame: Up to 5 observations per person, at baseline, 3 months, 6 months, 9 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Mg/dL per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Mg/dL per week | 0.459 (0.204) | 0.056 (0.043)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.322, Mixed Models Analysis

8. Primary Outcome: Health Knowledge Quiz Mean Total Score Change Per Week From Baseline to Termination
Description: Quiz of information covered during Lifestyle Balance classes, score range 0 - 30, worst to best. The study groups' average score changes per week were then compared.
Time Frame: Up to 4 observations per person,at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | 0.02 (0.01) | 0.01 (0.01)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.652, Mixed Models Analysis

9. Primary Outcome: Change in Mean Total Calories Consumed Per Week From Baseline to Termination
Description: Caloric intake assessed by dietitians using participant-recorded weekly food and exercise journals. The study groups' average change in total calories consumed per week were then compared.
Time Frame: Up to 19 observations per person, weekly for the first 2 months, then monthly for 10 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Calories per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Calories per week | -12.3 (12.37) | -6.8 (2.37)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.663, Mixed Models Analysis

10. Primary Outcome: Change in Mean Empty Calories Consumed Per Week From Baseline to Termination
Description: Caloric intake assessed by dietitians using participant-recorded weekly food and exercise journals. The study groups' average change in empty calories consumed per week were then compared.
Time Frame: Up to 19 observations per person, weekly for the first 2 months, then monthly for 10 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Calories per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Calories per week | -3.02 (11.79) | -4.53 (2.25)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.9, Mixed Models Analysis

11. Primary Outcome: Change in Mean Total Exercise Time Per Week From Baseline to Termination
Description: Minutes exercised assessed by dietitians using participant-recorded weekly food and exercise journals. The study groups' average change in total minutes exercised per week were then compared.
Time Frame: Up to 19 observations per person, weekly for the first 2 months, then monthly for 10 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Minutes per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Minutes per week | 0.84 (0.65) | 0.18 (0.47)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.415, Mixed Models Analysis

12. Primary Outcome: Mean University Rhode Island Change Assessment Scale (URICA) Total Score Change Per Week From Baseline to Termination
Description: Self-reported survey of respondents' feelings about changing their weight problem. Total score is also called the Readiness Score, ranging from -2 to +14 (worse to better), calculated by subtracting the mean from the precontemplation responses from the summation of the means of responses to contemplation, action, and the struggling to maintain items.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | -0.009 (0.006) | -0.006 (0.004)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.687, Mixed Models Analysis

13. Primary Outcome: WHO Quality of Life-BREF (WHOQOL-BREF) Mean Domain 1 Score Change Per Week From Baseline to Termination
Description: Self-reported survey of quality of life as related to respondents' physical health, score range 7-35, worst to best. The study groups' average subscore changes per week were then compared.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | 0.037 (0.016) | 0.013 (0.011)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.22, Mixed Models Analysis

14. Primary Outcome: WHO Quality of Life-BREF (WHOQOL-BREF) Mean Domain 2 Score Change Per Week From Baseline to Termination
Description: Self-reported survey of quality of life as related to respondents' psychological health, score range 6-30, worst to best. The study groups' average subscore changes per week were then compared.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | 0.027 (0.012) | -0.002 (0.009)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.059, Mixed Models Analysis

15. Primary Outcome: WHO Quality of Life-BREF (WHOQOL-BREF) Mean Domain 3 Score Change Per Week From Baseline to Termination
Description: Self-reported survey of quality of life as related to respondents' social relationships, score range 3-15, worst to best. The study groups' average subscore changes per week were then compared.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | 0.005 (0.011) | 0.008 (0.007)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.79, Mixed Models Analysis

16. Primary Outcome: WHO Quality of Life-BREF (WHOQOL-BREF) Mean Domain 4 Score Change Per Week From Baseline to Termination
Description: Self-reported survey of quality of life as related to respondents' environment, score range 8-40, worst to best. The study groups' average subscore changes per week were then compared.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | 0.03 (0.012) | 0 (0.011)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.146, Mixed Models Analysis

17. Primary Outcome: Brief Psychiatric Rating Scale (BPRS) Mean Total Score Change Per Week From Baseline to Termination
Description: Clinician-assessed symptom survey, score range 18 - 126, best to worst. The study groups' average score changes per week were then compared.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | -0.005 (0.001) | -0.002 (0.001)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p < .001, Mixed Models Analysis

18. Primary Outcome: Beck Anxiety Inventory (BAI) Mean Total Score Change Per Week From Baseline to Termination
Description: Self-reported symptom survey, score range 0 - 63, best to worst. The study groups' average score changes per week were then compared.
Time Frame: Up to 4 observations per person, at baseline, 2 months, 6 months, and 12 months.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Scores on a scale per week
Arm/Group | Usual Care | Lifestyle Balance
Number analyzed (Participants) | 42 | 62
Scores on a scale per week | -0.09 (0.05) | -0.11 (0.03)
Statistical Analysis 1: Comparison: Usual Care vs Lifestyle Balance; Test type: Superiority; p = 0.763, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: During 52-week period from participant randomization to termination.
Description: 17 participants in "Usual Care then Lifestyle Balance" group are included in both Usual Care and Lifestyle Balance arms, as they were exposed to both interventions. Events for these participants are reported per intervention, tallied under the intervention they were in at the time the event occurred.
Arm/Group | Usual Care | Lifestyle Balance
All-Cause Mortality (participants affected / at risk) | 1/59 | 2/79
Serious Adverse Events (participants affected / at risk) | 8/59 | 7/79
Other Adverse Events (participants affected / at risk) | 0/59 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=59) | Lifestyle Balance (N=79)
Death NOS (General disorders) | 1 (1) | 2 (2) — Caregiver-reported death of subject
Depression (Psychiatric disorders) | 0 (0) | 1 (1) — Hospitalization for recovery
Surgical and medical procedures - Other, specify (Cardiac disorders) | 1 (1) | 0 (0) — Pacemaker implantation
Surgical and medical procedures - Other, specify (Reproductive system and breast disorders) | 1 (1) | 0 (0) — Penile prosthesis implantation
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) — Hospitalization for recovery
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) — Hospitalization for recovery
Wound dehiscence (Eye disorders) | 0 (0) | 1 (1) — Hospitalization for recovery
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1) — Hospitalization for recovery
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Positive test for small cell neuroendocrine carcinoma
Agitation (Psychiatric disorders) | 1 (2) | 1 (2) — Hospitalization for recovery
Rectal pain (Gastrointestinal disorders) | 1 (3) | 0 (0) — Hospitalization for recovery
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Broken leg
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Hospitalization for recovery

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-02-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT01052714/Prot_SAP_000.pdf
  • Informed Consent Form (2011-10-13): https://cdn.clinicaltrials.gov/large-docs/14/NCT01052714/ICF_001.pdf